CLINICAL TRIAL: NCT03330145
Title: Risk Factors for Complicated Grief After a Death From Cancer or an Other Cause: A Longitudinal and Prospective Study Among Children and Their Parents
Brief Title: Complicated Grief Among Children After a Death From Cancer or Another Cause: A Longitudinal and Prospective Study (CAPS)
Acronym: CAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/15/7458
Record Dates: First submitted 2016-05-27; First posted 2017-11-06 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Grief
Keywords: Complicated Grief; Risk Factors; Cancer; Children
MeSH Terms: conditions — Neoplasms | interventions — Weights and Measures; Surveys and Questionnaires; Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- children who lost a parent to cancer (Experimental): Children will complete scales, questionnaires and inventory at 3 months post-loss and only 2 scales at 6 and 12 month post-loss
  Interventions: Behavioral: Scales, questionnaires and inventory
- children who lost a parent not to cancer (Active Comparator): Children will complete scales, questionnaires and inventory at 3 months post-loss and only 2 scales at 6 and 12 month post-loss
  Interventions: Behavioral: Scales, questionnaires and inventory

INTERVENTIONS:
Behavioral: Scales, questionnaires and inventory — Children will complete scales, questionnaires and inventory at 3 months post-loss and only 2 scales at 6 and 12 month post-loss
  Other Names: Inventory

SUMMARY:
The purpose of this study is to identify risk factors of Complicated Grief (CG) among children and adolescents who lost a parent to cancer or from an other cause.

DETAILED DESCRIPTION:
Although the intensity of the grief and life disruption usually subsides in the months following the loss of a loved one, approximately 7% of bereaved individuals will continue to experience persistent and intense grief-related symptoms associated with marked distress and functional impairment years after the death.

While several studies aimed to evaluate risk factors of CG among adults, little is known regarding CG among children and adolescents. Therefore, prospective research directly examining the impact of bereavement on post-loss psychiatric symptoms, including CG, post-traumatic-stress disorder (PTSD), depression, attentional and behavioral avoidance among children are needed. Improving our understanding of CG risk factors among children will help direct healthcare professionals' clinical attention toward screening and care of this underserved population.

Furthermore, identifying mechanisms explaining why cancer bereaved children may be at greater risk for persistent psychological distress and CG will inform the development of preventive, early intervention and treatment strategies.

Participants will be recruited to the Child and Adolescent grief counseling of the College Hospital of Toulouse as well as with the Team Regional Resource Pediatric Palliative Care "Enfant-Do". At 3, 6 and 12 months post-loss, children and their parent will be invited to complete questionnaires assessing peritraumatic dissociative experiences, peritraumatic distress, security attachment, symptoms of CG, symptoms of PTSD and attentional avoidance.

ELIGIBILITY:
Inclusion Criteria:

Children :

* Having lost a parent within the last 3 months
* Signed consent form from the parent
* To have health care coverage by the French social security

Parents :

* Signed consent form
* Having lost mother or father of the child within the last 3 months

Exclusion Criteria:

Children:

* Both parents are dead
* Medical disease
* Ongoing legal procedure regarding the death

Parents :

* Decline to take part to the study
* Mental retardation or schizophrenia
* Ongoing legal procedure regarding the death

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Inventory of Complicated Grief | 6 months post-loss
  Complicated Grief symptoms at 6 months post-loss among children aged from 6 to 17 years Measured by the Inventory of Complicated Grief

SECONDARY OUTCOMES:
Inventory of Complicated Grief for Evaluation of paths of grief symptoms developement | At 3 and 12 months post-loss
  Analysed symptoms and divided subject between 4 groups according to their symptoms.
  Group 1 : High levels of grief symptoms at 3 months wich will decrease at 12 months Group 2 : Low levels of grief symptoms at 3 months wich will stay low at 12 months Group 3 : High levels of grief symptoms at 3 months wich will stay high at 12 months Group 4 : Low levels of grief symptoms at 3 months wich will increase at 12 months
Influence of grief symptoms of the parent staying in life | At 3 months and 12 months post-loss
  Evaluation of the influence of grief symptoms of the parent staying in life on the level of complicated grief symptoms development (i) One group of children will have high levels of grief symptoms at T0 which will decrease over the time.
  (ii) One group will have low levels of grief symptoms at T0 which will remain low over the time.
  (iii) One group will have high levels of grief symptoms at T0 which will remain high over the time.
  (iiii) One group will have low levels of grief symptoms at T0 which will increase over the time.
Evaluation of the impact of the cause of parents death (cancer or other cause) on complicated grief symptoms development. | At 6 and 12 months post-loss
  Questionnaire will be used to measure these symptoms : Inventory of Complicated Grief
Evaluation of the impact of the cause of parents death (cancer or other cause) on post-traumatic stress developement. | At 6 and 12 months post-loss
  Questionnaires will be used to measure these symptoms : Peritraumatic Dissociative Experiences Questionnaire and Peritraumatic Distress Inventory
Evaluation of the impact of the cause of parents death (cancer or other cause) on depression developement. | At 6 and 12 months post-loss
  Questionnaire will be used to measure these symptoms : Children Depression Inventory
Determined if early factors could explain differences of symptoms of complicated grief between the cause of death of the parent (cancer or another cause) | At 3 months post-loss
  Questionnaire will be used to measure these symptoms : Inventory of Complicated Grief
Determined if early factors could explain differences of symptoms of post-traumatic stress developement between the cause of death of the parent (cancer or another cause) | At 3 months post-loss
  Questionnaire will be used to measure these symptoms : Peritraumatic Dissociative Experiences Questionnaire and Peritraumatic Distress Inventory
Determined if early factors could explain differences of symptoms of depression developement between the cause of death of the parent (cancer or another cause) | At 3 months post-loss
  Questionnaire will be used to measure these symptoms : Children Depression Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe RAYNAUD, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Psychiatrie de l'enfant et de l'adolescent, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Revet A, Suc A, Auriol F, Djelantik AAAMJ, Raynaud JP, Bui E. Peritraumatic distress predicts prolonged grief disorder symptom severity after the death of a parent in children and adolescents. Eur J Psychotraumatol. 2021 Jun 28;12(1):1936916. doi: 10.1080/20008198.2021.1936916. eCollection 2021. PMID 34249245